CLINICAL TRIAL: NCT03258853
Title: Feasibility of Outpatient Automated Blood Glucose Control With the iLet Bionic Pancreas for Treatment of Cystic Fibrosis Related Diabetes
Brief Title: Feasibility of Outpatient Closed Loop Control With the iLet Bionic Pancreas in Cystic Fibrosis Related Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beta Bionics, Inc. (Industry)
Responsible Party: Principal Investigator, Melissa Susan Putman, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020P003452
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis-related Diabetes
Keywords: cystic fibrosis; insulin; glucagon; continuous glucose monitor; bionic pancreas
MeSH Terms: conditions — Cystic Fibrosis; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Usual Care (Active Comparator): Usual Care diabetes management: Patients will manage their diabetes using standard of care for diabetes as per their typical regimen including use of an insulin pump or injectable insulin. Usual care arm for 14 days. Patients will wear a continuous glucose monitor (CGM) during this arm
  Interventions: Other: Usual Care
- Insulin only bionic pancreas (Experimental): Insulin Only Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin using a continuous glucose monitoring (CGM) device, for 14 days.
  Interventions: Device: Bionic Pancreas

INTERVENTIONS:
Device: Bionic Pancreas — Bionic pancreas system: The bionic pancreas is an autonomous, self-learning system that requires only the subject's weight for initialization, and then autonomously adapts insulin dosing to maintain glycemic control. The bionic pancreas uses continuous glucose monitoring as input to the controller. The bionic pancreas can be used in a bi-hormonal configuration, administering both insulin and glucagon as well as an insulin only setting.
  Arms: Insulin only bionic pancreas
Other: Usual Care — Subjects will remain on home insulin regimen (either insulin pump or injectable insulin). Subjects in usual care will wear a study CGM even if in typical care does not include CGM use.
  Arms: Usual Care

SUMMARY:
The current study is designed to test the feasibility of the a wearable bionic pancreas system that automatically delivers insulin and glucagon can provide superior regulation of glycemia versus usual care for adults and children with cystic fibrosis related diabetes.

ELIGIBILITY:
Inclusion criteria

* Age >/= 10 years and have had a diagnosis of cystic fibrosis related diabetes (CFRD) managed using either an insulin pump or multiple daily injections (MDI).
* Mean continuous glucose monitoring (CGM) glucose >/=125 mg/dl as determined by the participant's personal CGM 30-day download if CGM is used as part of their usual care. If the participant does not use CGM, hemoglobin A1c >/= 6% within the last 6-months from available medical records will be required.
* Minimum insulin requirement of >/=0.1u/kg/day. To ensure that participants with a wide range of insulin requirements are included, participants whose insulin requirement is <0.3u/kg/day will be limited to approximately 1/3 of the enrolled >/=18 year old adult cohort.
* Willing to wear iLet infusion sets and one Dexcom CGM sensor and change sets at least every other day in the iLet arm
* Assent will be obtained for patients <18 of age

Exclusion criteria

* Diabetes from etiologies other than CFRD
* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory, unable to speak and read English)
* Current participation in another clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the participant
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the next 3-months, or sexually active without use of contraception

  o Participants must use acceptable contraception for the two weeks prior to the study, throughout the study and for the two weeks following the study.
* History of hypoglycemic seizures (grand-mal) or coma in the last year
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
* Unable to avoid hydroxyurea for duration of study (interferes with accuracy of Dexcom G6 CGM)
* Unable to avoid taking higher than the maximum dose of acetaminophen from all sources for the duration of the study (interferes with accuracy of Dexcom G6 CGM)

  * Adult: 1 g every 6 hours, up to 4 g every 24 hours
  * Pediatric: 75 mg/kg/day in up to 5 doses, not to exceed 4000 mg/day
* Have started or stopped a cystic fibrosis transmembrane conductance regulator (CFTR) modulator in the past 4 weeks.
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* Use of oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, DPP-4 inhibitors, SGLT-2 inhibitors) or non-insulin injectable (GLP-1 agonists, amylin) anti-diabetic medications
* History of lung or liver transplant
* Anticipated lung transplant (on transplant list)
* No acute pulmonary exacerbation or hospitalizations within the past 4 weeks or treatment with IV antibiotics in the past 4 weeks.
* Any factors that, in the opinion of the principal investigator would interfere with the safe completion of the study
* History of severe liver disease, including cirrhosis or portal hypertension
* Presence of a medical condition or use of a medication that, in the judgment of the investigator, could compromise the results of the study or the safety of the participant. Conditions to be considered by the investigator may include the following:

  * Current alcohol abuse (intake averaging >3 drinks daily in last 30 days) or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
  * Unwilling or unable to refrain from drinking more than 2 drinks in an hour or more than 4 drinks in a day during the trial
  * Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of beta blockers will be allowed as long as the dose is stable and the participant does not meet the criteria for hypoglycemia unawareness while taking that stable dose, but use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
  * Renal failure requiring dialysis
  * Any known history of coronary artery disease including, but not limited to, history of myocardial infarction, stress test showing ischemia, history of angina, or history of intervention such as coronary artery bypass grafting, percutaneous coronary intervention, or enzymatic lysis of a presumed coronary occlusion)
  * Congestive heart failure (established history of CHF, lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea) oHistory of TIA or stroke
  * Seizure disorder, history of any non-hypoglycemic seizure within the last two years, or ongoing treatment with anticonvulsants
  * History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Putman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De identified glucose data and microbiome data will be shared with research collaborators.
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 2021 and June 2022
Pre-assignment Details: 30 adults were consented and screened for study participation. Of these, 3 did not meet inclusion criteria, 3 declined to participate, and 2 were lost to follow-up prior to randomization. The remaining 22 subjects were randomized. 2 subjects were assigned to a study arm but withdrew prior to any study procedures. No baseline or outcome data were collected in these 2 subjects, and they were excluded from all analyses. The remaining 20 subjects completed the study and are included in the analyses.
Groups:
- Usual Care First, Then Insulin Only Bionic Pancreas: Usual Care diabetes management: Patients will manage their diabetes using standard of care for diabetes as per their typical regimen including use of an insulin pump or injectable insulin. Usual care arm for 14 days. Patients will wear a continuous glucose monitor (CGM) during this arm
  Usual Care: Subjects will remain on home insulin regimen (either insulin pump or injectable insulin). Subjects in usual care will wear a study CGM even if in typical care does not include CGM use.
  After completing 14 days of Usual Care, participants then crossed over to the insulin only bionic pancreas for another 14 days.
  Insulin Only Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin using a continuous glucose monitoring (CGM) device, for 14 days.
  Bionic Pancreas: Bionic pancreas system: The bionic pancreas is an autonomous, self-learning system that requires only the subject's weight for initialization, and then autonomously adapts insulin dosing to maintain glycemic control. The bionic pancreas uses continuous glucose monitoring as input to the controller. The bionic pancreas can be used in a bi-hormonal configuration, administering both insulin and glucagon as well as an insulin only setting.
- Insulin Only Bionic Pancreas First, Then Usual Care: Insulin Only Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin using a continuous glucose monitoring (CGM) device, for 14 days.
  Bionic Pancreas: Bionic pancreas system: The bionic pancreas is an autonomous, self-learning system that requires only the subject's weight for initialization, and then autonomously adapts insulin dosing to maintain glycemic control. The bionic pancreas uses continuous glucose monitoring as input to the controller. The bionic pancreas can be used in a bi-hormonal configuration, administering both insulin and glucagon as well as an insulin only setting.
  After completing 14 days of the insulin only bionic pancreas, participants then crossed over to Usual Care for another 14 days:
  Usual Care diabetes management: Patients will manage their diabetes using standard of care for diabetes as per their typical regimen including use of an insulin pump or injectable insulin. Usual care arm for 14 days. Patients will wear a continuous glucose monitor (CGM) during this arm
  Usual Care: Subjects will remain on home insulin regimen (either insulin pump or injectable insulin). Subjects in usual care will wear a study CGM even if in typical care does not include CGM use.
Period: First Intervention (14 Days)
Arm/Group | Usual Care First, Then Insulin Only Bionic Pancreas | Insulin Only Bionic Pancreas First, Then Usual Care
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention (14 Days)
Arm/Group | Usual Care First, Then Insulin Only Bionic Pancreas | Insulin Only Bionic Pancreas First, Then Usual Care
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care First, Then Insulin Only Bionic Pancreas: Usual Care diabetes management: Patients will manage their diabetes using standard of care for diabetes as per their typical regimen including use of an insulin pump or injectable insulin. Usual care arm for 14 days. Patients will wear a continuous glucose monitor (CGM) during this arm
  Usual Care: Subjects will remain on home insulin regimen (either insulin pump or injectable insulin). Subjects in usual care will wear a study CGM even if in typical care does not include CGM use.
  After 14 days of Usual Care, participants then crossed over to the Insulin only bionic pancreas arm for anther 14 days.
  Insulin Only Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin using a continuous glucose monitoring (CGM) device, for 14 days.
  Bionic Pancreas: Bionic pancreas system: The bionic pancreas is an autonomous, self-learning system that requires only the subject's weight for initialization, and then autonomously adapts insulin dosing to maintain glycemic control. The bionic pancreas uses continuous glucose monitoring as input to the controller. The bionic pancreas can be used in a bi-hormonal configuration, administering both insulin and glucagon as well as an insulin only setting.
- Insulin Only Bionic Pancreas First, Then Usual Care: Insulin Only Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin using a continuous glucose monitoring (CGM) device, for 14 days.
  Bionic Pancreas: Bionic pancreas system: The bionic pancreas is an autonomous, self-learning system that requires only the subject's weight for initialization, and then autonomously adapts insulin dosing to maintain glycemic control. The bionic pancreas uses continuous glucose monitoring as input to the controller. The bionic pancreas can be used in a bi-hormonal configuration, administering both insulin and glucagon as well as an insulin only setting.
  After 14 days of the insulin only bionic pancreas, participants then crossed over to the usual care arm for another 14 days.
  Usual Care diabetes management: Patients will manage their diabetes using standard of care for diabetes as per their typical regimen including use of an insulin pump or injectable insulin. Usual care arm for 14 days. Patients will wear a continuous glucose monitor (CGM) during this arm
  Usual Care: Subjects will remain on home insulin regimen (either insulin pump or injectable insulin). Subjects in usual care will wear a study CGM even if in typical care does not include CGM use.
- Total: Total of all reporting groups
Arm/Group | Usual Care First, Then Insulin Only Bionic Pancreas | Insulin Only Bionic Pancreas First, Then Usual Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (17) | 39 (10) | 40 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 10 | 18
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (3.2) | 23.8 (4.9) | 23.7 (3.5)
HbA1c [Mean (Standard Deviation); unit: % of glycated hemoglobin] | 8.0 (1.5) | 6.2 (2.7) | 7.4 (1.6)
Mean CGM glucose [Mean (Standard Deviation); unit: mg/dL] | 173 (35) | 163 (25) | 167 (29)
Cystic fibrosis related diabetes (CFRD) duration [Mean (Standard Deviation); unit: years] | 13 (9) | 17 (10) | 15 (10)
Insulin Total Daily Dose [Mean (Standard Deviation); unit: units/kg/day] | 0.62 (0.26) | 0.46 (0.30) | 0.54 (0.29)
Percent predicted forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: % of predicted] | 76 (26) | 65 (21) | 70 (24)
Pancreatic insufficiency [Count of Participants; unit: Participants] | 10 | 10 | 20
Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Modulator Use [Count of Participants; unit: Participants] | 7 | 10 | 17
Continuous glucose monitor (CGM) Use [Count of Participants; unit: Participants] | 8 | 10 | 18
Multiple Daily Injection Use [Count of Participants; unit: Participants] | 7 | 3 | 10
Insulin Pump Use [Count of Participants; unit: Participants] | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Glucose Target Range (70-180 mg/dl) as Determined by Continuous Glucose Monitor (CGM) on Days 3-14
Description: Percentage of time spent with CGM glucose values between 70 and 180 mg/dl
Time Frame: Days 3-14
Population: This was a random-order cross-over design clinical trial. Each participant completed each study arm.
Measure: Mean (Standard Deviation); unit: percentage of time spent in target range
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
percentage of time spent in target range | 63 (22) | 75 (11)
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.001, paired 2-sided t-test

2. Secondary Outcome: Percentage of Time Spent With CGM Glucose: < 54 mg/dl
Description: Percentage of time spent with CGM glucose in this range
Time Frame: Days 3-14
Measure: Median (Inter-Quartile Range); unit: percentage of time spent <54mg/dL
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
percentage of time spent <54mg/dL | 0.36 [0 to 0.82] | 0.27 [0.06 to 0.76]
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 1.0, Wilcoxon signed rank test — Secondary outcomes were adjusted for multiple comparisons

3. Secondary Outcome: Mean CGM Glucose
Description: Average CGM glucose
Time Frame: Days 3-14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
mg/dL | 171 (45) | 150 (19)
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.04, paired 2-sided t-test — Secondary outcomes are adjusted for multiple comparisons

4. Secondary Outcome: Percentage of Time Spent With CGM Glucose < 70 mg/dl
Description: Percent of time the participant spent with CGM glucose in this range
Time Frame: Days 3-14
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
percentage of time | 1.5 [0.13 to 3.5] | 1.7 [1.0 to 2.5]
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 1.0, Wicoxon signed rank test — Adjusted for multiple comparisons

5. Secondary Outcome: Percentage of Time Spent With CGM Glucose >180 mg/dL
Description: The percent of time the participant spent with CGM glucose in this range
Time Frame: Days 3-14
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
percentage of time | 31 [17 to 52] | 18 [14 to 31]
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.014, Wilcoxon signed rank test — Adjusted for multiple comparisons

6. Secondary Outcome: Percentage of Time Spent With CGM Glucose > 250mg/dL
Description: The percent of time the participant spent with CGM glucose in this range
Time Frame: Days 3-14
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
percentage of time | 10 [2.5 to 22] | 3.9 [2.0 to 9.7]
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.014, Wilcoxon signed rank test — Adjusted for multiple comparisons

7. Secondary Outcome: Standard Deviation
Description: Standard deviation of participants' mean CGM glucose
Time Frame: Days 3-14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
mg/dL | 60 (16) | 54 (15)
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.14, Wilcoxon signed rank test — Adjusted for multiple comparisons

8. Secondary Outcome: Coefficient of Variation
Description: Coefficient of variation of CGM glucose values
Time Frame: Days 3-14
Measure: Mean (Standard Deviation); unit: percentage of variability
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
percentage of variability | 35 (6) | 35 (6)
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 1.0, Wilcoxon signed rank test — Adjusted for multiple comparisons

9. Secondary Outcome: Number of Episodes of Self-reported Symptomatic Hypoglycemia
Description: Number of episodes subjects reported experiencing symptoms of low blood sugar (hypoglycemia)
Time Frame: Days 3-14
Measure: Median (Inter-Quartile Range); unit: Episodes
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
Episodes | 0.4 [0 to 0.8] | 0.7 [0.4 to 1.2]
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.01, Wilcoxon signed rank test

10. Secondary Outcome: Number of Subjects With Mean CGMG <154 mg/dl
Description: Number of subjects who achieve a mean CGM glucose < 154 mg/dl, which is the estimated average glucose for a hemoglobin A1c of 7% (ADA goal for therapy)
Time Frame: Days 3-14
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
Participants | 9 | 12
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.08, McNemar

11. Secondary Outcome: Number of Subjects With Percentage of Time < 54 mg/dl < 1%
Description: Number of subjects who have less than 1% percent of CGM glucose values < 54 mg/dl
Time Frame: Days 3-14
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
Participants | 17 | 16
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.56, McNemar

12. Secondary Outcome: Number of Subjects With Percentage of Time < 54 mg/dl < 1% and Mean CGM Glucose < or Equal to 154 mg/dl
Description: Number of subjects who have less than 1% percent of CGM glucose values < 54 mg/dl and also have a mean CGM glucose that is less than or equal to 154 mg/dl
Time Frame: Days 3-14
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
Participants | 7 | 8
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.56, McNemar

13. Secondary Outcome: Number of Subjects With Time in Range (70-180 mg/dl) of 70% or Greater
Description: Number of subjects who have 70% percent or more of their CGM glucose values between 70 and 180 mg/dl
Time Frame: Days 3-14
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 20 | 20
Participants | 9 | 11
Statistical Analysis 1: Comparison: Usual Care vs Insulin Only Bionic Pancreas; Test type: Superiority; p = 0.15, McNemar

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after screening and enrollment until the participant completed both arms of the trial, each 14 days in duration.
Arm/Group | Usual Care | Insulin Only Bionic Pancreas
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=20) | Insulin Only Bionic Pancreas (N=20)
Hyperglycemia without ketosis (Endocrine disorders) | 0 (0) | 5 (6)
Hyperglycemia with ketosis (Endocrine disorders) | 1 (2) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycemia unawareness (Endocrine disorders) | 1 (1) | 0 (0)
Pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT03258853/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT03258853/ICF_001.pdf